CLINICAL TRIAL: NCT01037699
Title: Luteinizing Hormone (LH) Supplementation in Gonadotropin-releasing Hormone (GnRH) Antagonist Cycles
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Instituto Valenciano de Infertilidad, IVI VALENCIA (Other)
Responsible Party: Dr. Ernesto Bosch, IVI Valencia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0502-C-M05-EB
Record Dates: First submitted 2009-12-21; First posted 2009-12-23 (Estimated); Last update posted 2009-12-23 (Estimated); Status verified 2009-12

CONDITIONS: Ovarian Stimulation
Keywords: Ovarian stimulation; In Vitro Fertilization; Luteinizing Hormone; GnRH antagonist; Implantation rate in infertile patients undergoing In vitro fertilization and embryo transfer.

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- FSH YOUNGER (Active Comparator)
  Interventions: Drug: rFSH: Follicle Stimulating Hormone
- FSH OLDER (Active Comparator)
  Interventions: Drug: rFSH: Follicle Stimulating Hormone
- FSH LH YOUNGER (Recombinant Luteotrophin alfa) (Experimental)
  Interventions: Drug: rFSH: Follicle Stimulating Hormone and rLH: Luteinizing Hormone (Recombinant Luteotrophin alfa)
- FSH LH OLDER (Experimental)
  Interventions: Drug: rFSH: Follicle Stimulating Hormone and rLH: Luteinizing Hormone (Recombinant Luteotrophin alfa)

INTERVENTIONS:
Drug: rFSH: Follicle Stimulating Hormone
  Arms: FSH YOUNGER
Drug: rFSH: Follicle Stimulating Hormone
  Arms: FSH OLDER
Drug: rFSH: Follicle Stimulating Hormone and rLH: Luteinizing Hormone (Recombinant Luteotrophin alfa)
  Arms: FSH LH YOUNGER (Recombinant Luteotrophin alfa)
Drug: rFSH: Follicle Stimulating Hormone and rLH: Luteinizing Hormone (Recombinant Luteotrophin alfa)
  Arms: FSH LH OLDER

SUMMARY:
To analyse the impact on cycle outcome of LH supplementation in ovarian stimulation controlled with a GnRH antagonist in two ages groups: patients upto 35 years old, and patients aged between 36 and 39 years old.

DETAILED DESCRIPTION:
All patients received an oral contraceptive pill with 0.030 mg of ethinyl-estradiol and 3.0 mg of drospirenone the cycle prior to ovarian stimulation. On the second day of menstruation, patients started ovarian stimulation as follows:

Patients < 36: 225 IU/day of recombinant FSH (FSH alone group) or 150 IU of rFSH and 75 IU of rLH/day (FSH+LH group) for 5 days. On day 6, a 0.25 mg/day dose of the GnRH antagonist Cetrorelix is added until the day of rCG administration.

Patients 36-39: Initial dose of 300 IU of rFSH /day (FSH alone group)) or 225 IU of rFSH and 75 IU of rLH/day (FSH + LH group) for 5 days. On day 6, a 0.25 mg/day dose of the GnRH antagonist Cetrorelix is added until the day of rCG administration.

A maximum of 3 embryos were transferred on day 3 of embryo development.

ELIGIBILITY:
Inclusion Criteria:

* 1st-2nd IVF cycle.
* Age until 39 years old
* BMI: 18-29.9.
* Basal FSH < 12 IU/L

Exclusion Criteria:

* LH:FSH > 2 (PCO)
* Low response background (< 5 oocytes)
* Endometrioma
* Recurrent pregnancy loss
* Any preimplantational genetic diagnosis indication
* Any systemic, metabolic or endocrinological disorder.

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 720 (Actual)
Dates: Start 2005-01; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Implantation rate | 4 weeks after embryo transfer

CONTACTS AND LOCATIONS:
Overall Officials: Ernesto Bosch, MDPhD, Principal Investigator — IVI Valencia
Locations (1):
- IVI Valencia, Valencia, Valencia, Spain